CLINICAL TRIAL: NCT00642707
Title: A Phase 2a, Randomized, Double-blind, Placebo Controlled Study of PRO 140 by Subcutaneous Administration in Adult Subjects With Human Immunodeficiency Virus Type 1 Infection
Brief Title: Study of PRO 140 by Subcutaneous Administration in Adult Subjects With HIV -1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO 140 2101
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: HIV -1 Infection; HIV Infections
Keywords: HIV; Treatment Naïve
MeSH Terms: conditions — HIV Infections | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator): PRO 140 for three single SC doses: Days 1, 8, and 15
  Interventions: Drug: PRO 140 (humanized monoclonal antibody to CCR5)
- Arm 2 (Active Comparator): PRO 140 for three single SC doses: Days 1, 8 and 15
  Interventions: Drug: PRO 140 (humanized monoclonal antibody to CCR5)
- Arm 3 (Active Comparator): PRO 140 for two single SC doses: Days 1 and 15 plus one SC dose of PBO at Day 8
  Interventions: Drug: PRO 140 (humanized monoclonal antibody to CCR5)
- Arm 4 (Placebo Comparator): PBO for three single SC doses: Days 1, 8 and 15
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: PRO 140 (humanized monoclonal antibody to CCR5)
  Arms: Arm 1; Arm 2; Arm 3
Drug: Placebo Comparator
  Arms: Arm 4

SUMMARY:
The purpose of this study is:

1. To assess the antiviral activity of PRO 140
2. To assess the safety and tolerability of PRO 140
3. To generate additional PK, PD and safety data of PRO 140

ELIGIBILITY:
Inclusion Criteria:

1. Males & females, age ≥ 18 years (or minimum adult age as determined by local regulatory authorities)
2. Screening plasma HIV-1 RNA ≥ 5,000 copies/mL
3. CD4+ lymphocyte cell count ≥ 300 cells/mm3 and no documented count < or = 250 cells/mm3
4. Has not taken any antiretroviral therapy (ART) w/in 12 wks of Early Screening Visit
5. Exclusive CCR5-tropic virus as determined by Trofile™ Assay at Early Screening Visit
6. Clinically normal or "not clinically significant (NCS)" resting electrocardiogram
7. Women of reproductive potential must have a negative serum pregnancy test at Late Screening Visit & a negative urine pregnancy test w/in 72 hrs prior to first dose of study medication, & be non-lactating. Male & female subjects must agree not to participate in a conception process from Early Screening Visit through Day 59.

Exclusion Criteria:

1. CXCR4 tropic virus or dual/mixed tropic (R5X4) virus determined by the Trofile™ Assay.
2. Females who are pregnant, lactating or breastfeeding, or who plan to become pregnant during the study.
3. History of active hepatitis within the previous 24 wks
4. Prior use of any entry, attachment, CCR5 co-receptor or fusion inhibitor, including PRO 140, experimental or approved.
5. Any immunization or vaccination (including influenza vaccine) within 30 days prior to administration of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Morris, MD, PhD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States

REFERENCES:
- [Derived] Jacobson JM, Thompson MA, Lalezari JP, Saag MS, Zingman BS, D'Ambrosio P, Stambler N, Rotshteyn Y, Marozsan AJ, Maddon PJ, Morris SA, Olson WC. Anti-HIV-1 activity of weekly or biweekly treatment with subcutaneous PRO 140, a CCR5 monoclonal antibody. J Infect Dis. 2010 May 15;201(10):1481-7. doi: 10.1086/652190. PMID 20377413
- See also: Related Info — http://www.progenics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started March 2008 and ended November 2008
Pre-assignment Details: There was a screening period of up to 12 weeks. Subjects had to be infected with CCR5-tropic human immunodeficiency virus type 1 (HIV-1)or they were excluded from the study.
Groups:
- Arm 1: PRO 140 - 162 mg for three single SC doses: Days 1, 8, and 15
- Arm 2: PRO 140 - 324 mg for three single SC doses: Days 1, 8 and 15
- Arm 3: PRO 140 - 324 mg for two single SC doses: Days 1 and 15 plus one SC dose of placebo at Day 8
- Arm 4: Placebo for three single SC doses: Days 1, 8 and 15
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 11 | 11 | 12 | 10
Completed | 10 | 11 | 12 | 8
Not Completed | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 11 | 11 | 12 | 10 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 12 | 10 | 44
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (5.13) | 41.9 (5.46) | 46.4 (8.18) | 42.4 (7.44) | 42.4 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 10 | 10 | 11 | 9 | 40
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 12 | 10 | 44

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change in Viral Load Following Initiation of Treatment (Viral Load is Defined as HIV-1 Copies/mL and Expressed as log10 Copies/mL).
Description: The primary end point was the maximum change from baseline in viral load following initiation of treatment, defined as HIV-1 copies/mL, measured by the Roche Amplicor HIV-1 Monitor UltraSensitive™ Test (lower limit of detection [LLD] = 48 copies/mL).
Time Frame: 59 days
Population: All randomized subjects who received one dose of study drug were considered intent-to-treat (ITT) subjects and were analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: Log10copies/HIV-1 RNA/mL
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 11 | 11 | 12 | 10
Log10copies/HIV-1 RNA/mL | -0.99 (0.558) | -1.65 (0.571) | -1.37 (0.891) | -0.23 (0.285)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 3/12 | 0/10
Other Adverse Events (participants affected / at risk) | 9/11 | 10/11 | 11/12 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm 1 (N=11) | Arm 2 (N=11) | Arm 3 (N=12) | Arm 4 (N=10)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1/1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1/1 (1) | 0 (0)
Anal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1/1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm 1 (N=11) | Arm 2 (N=11) | Arm 3 (N=12) | Arm 4 (N=10)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Perianal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site induration (General disorders) | 1 (3) | 2 (5) | 3 (5) | 0 (0)
Infusion site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abcess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syphillis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Chemical poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex serology positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Anal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile discharge (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Because the study is a multicenter study, the PI(s) can only publish after the aggregate results of all investigators and institutions participating in the study have been published, and the proposed publication is reviewed by Progenics. In the event that Progenics does not publish the results of the study within eighteen months from availability of final study analysis, the PI can publish provided that the proposed publication is reviewed by Progenics.